CLINICAL TRIAL: NCT06874855
Title: Lemborexant in Delayed Sleep Phase Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eisai Co., Ltd. (Industry); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-38738
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Delayed Sleep Phase Syndrome
Keywords: Delayed Sleep Phase Syndrome; Syndrome; Lemborexant
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Syndrome | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: To evaluate whether Lemborexant is more effective than placebo in shortening sleep onset latency in patients with delayed sleep phase syndrome (both type 1 and type 2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Patients receive placebo to match Lemborexant for 14 days
  Interventions: Drug: Placebo
- Lemborexant (Active Comparator): Patients receive Lemborexant 5mg for 7 days and may be dose adjusted to 10mg. Patients continue to take Lemborexant 5mg or 10mg for an additional 7 days
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — Lemborexant tablet administered orally once daily
  Other Names: dayvigo
  Arms: Lemborexant
Drug: Placebo — Placebo to match Lemborexant tablet administered orally once daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether Lemborexant is more effective than placebo in shortening sleep onset latency in patients with delayed sleep phase syndrome (both type 1 and type 2). This will be tracked using sleep logs as well as actigraphy.

In this 2-year study, the investigators will examine if Lemborexant administered 5-10 mg nightly taken at desired bedtime (at least 2 hours prior to self-reported sleep onset habitual time) can improve the symptoms of Delayed Sleep Phase Syndrome.

DETAILED DESCRIPTION:
Delayed sleep phase syndrome (DSPS) is a disorder in which a person's sleep is delayed by two hours or more beyond what is considered an acceptable or conventional bedtime. The delayed sleep then causes difficulty in being able to wake up at the desired time. In DSPS, bedtime is shifted later than the general population such that individuals have difficulty getting enough sleep to meet their sleep need before they have to get up for their daytime obligations (work, school, childcare, etc.). As a result, patients experience daytime impairment including daytime sleepiness and cognitive impairment. DSPS, if maintained in adulthood is associated with numerous deleterious health effects, although causality is not well established. The prevalence of this condition is approximately 7-16% among adolescents and young adults.

ELIGIBILITY:
Inclusion Criteria:

- Participants will be required to be 18 years of age or older and have delayed sleep phase syndrome (DSPS). Questionnaires will be used to identify potential confounders and to confirm a potential diagnosis of DSPS based on ICSD3 criteria: a) Sleep is delayed by two hours or more beyond what is considered an acceptable or conventional bedtime for the subject (their desired bedtime). b) Subjects not able to fall asleep if trying to sleep before the later bedtime; c) This is interfering with their wishes/having a social impact. Concomitant medications will be allowed, though dosages will be required to remain fixed throughout participation in the study. The participant also needs to be willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

* Clinically significant depression (PHQ-9 score of 10 or more), anxiety disorder (GAD- 7 score of 10 or more), substance use disorder, any other sleep disorder, or any medical disorder/therapy that could interfere with the trial
* Use of medications with significant effects on sleep-wake function (insomnia therapies, stimulants)- unless they are discontinued at least 5 half-lives prior to study participation. Non-sedative antidepressants or SSRI will be allowed if at a stable dose in the absence of concomitant severe depression or severe anxiety.
* Use of CYP3A inhibitors and CYP3A inducers, at least 1 week (or five half-lives, whichever is longer) prior to the first day of the baseline phase.
* Pregnancy (verified by urine pregnancy test on visits 1, 2, and 3) or plan to become pregnant in the next 3 months or currently breastfeeding.
* Shift workers or subjects working unusual hours.
* Transmeridian travel across more than 3 time zones 4 weeks prior to the screening phase.
* Transmeridian travel across more than 2 time zones during this trial (including the screening phase).
* Having a positive drug test or being unwilling to refrain from using illegal drugs or marijuana during this trial.
* Any clinically abnormal symptom or organ impairment found by medical history at Screening or Baseline and physical examinations, vital signs, or laboratory test results that require medical treatment.
* Impaired liver function (values for enzymes aspartate transaminase (AST) and alanine transaminase (ALT) > 1.5 times the Upper Limit of Normal).
* Known to be human immunodeficiency virus positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in actigraphy sleep latency onset | From 2 weeks prior to randomization to 4 weeks post randomization
  Sleep latency is the time from laying down until falling asleep. Actigraphy data obtained using Axivity- AX6.

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale (ESS) | From randomization to 4 weeks post randomization
  This is a scale to evaluate daytime sleepiness. Range from 0 to 24 points (higher scores mean more sleepiness).
Change in Karolinska Sleepiness Scale (KSS) | From randomization to 4 weeks post randomization
  Self-report for daytime sleepiness with 1 being extremely alert and 10 being extremely sleepy, can't keep awake.
Change in sleep diary derived sleep onset latency | From 2 weeks prior to randomization to 4 weeks post randomization
  Sleep latency is the time from laying down until falling asleep as estimated by patient in dairy.
Sleep Regularity Index | From 2 weeks prior to randomization to 4 weeks post randomization
  Sleep Regularity Index is defined as the percentage probability of a person being asleep (or awake) at any two time points 24 hours apart. Actigraphy data obtained using Axivity- AX6.
Change in actigraphy derived total sleep time | From 2 weeks prior to randomization to 4 weeks post randomization
  Actigraphy data obtained using Axivity- AX6.
Change in sleep diary derived total sleep time. | From 2 weeks prior to randomization to 4 weeks post randomization
  Estimated by patient in dairy.
Change in mean actigraphy derived wake time | From 2 weeks prior to randomization to 4 weeks post randomization
  Wake time is total time awake over night after sleep onset. Actigraphy data obtained using Axivity- AX6.
Change in mean sleep diary derived wake time | From 2 weeks prior to randomization to 4 weeks post randomization
  Wake time is total time awake over night after sleep onset as estimated by patient in dairy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krystal, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared only with collaborators at Stanford University who are mirroring this study and recruiting half of the required participants and with Eisai Inc Ltd, the study sponsor that is providing the drug of investigation. Individuals will be assigned a unique coded identifier to limit risk of privacy loss
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD from enrolled participants will be available to collaborators for the duration of the study (Mar 2023 - May 2027 (anticipated) until the study has ended.
Access Criteria: Collaborator Emmanuel Mignot from Stanford University and study sponsor Eisai will be able to access the data as participants from UCSF and Stanford will be combined for the overall data analyses

REFERENCES:
- [Background] Duffy JF, Dijk DJ, Hall EF, Czeisler CA. Relationship of endogenous circadian melatonin and temperature rhythms to self-reported preference for morning or evening activity in young and older people. J Investig Med. 1999 Mar;47(3):141-50. PMID 10198570
- [Background] Micic G, Richardson C, Cain N, Reynolds C, Bartel K, Maddock B, Gradisar M. Readiness to change and commitment as predictors of therapy compliance in adolescents with Delayed Sleep-Wake Phase Disorder. Sleep Med. 2019 Mar;55:48-55. doi: 10.1016/j.sleep.2018.12.002. Epub 2018 Dec 14. PMID 30763869
- [Background] Zeitzer JM, Joyce DS, McBean A, Quevedo YL, Hernandez B, Holty JE. Effect of Suvorexant vs Placebo on Total Daytime Sleep Hours in Shift Workers: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206614. doi: 10.1001/jamanetworkopen.2020.6614. PMID 32484552
- [Background] Zeitzer JM, Buckmaster CL, Lyons DM, Mignot E. Increasing length of wakefulness and modulation of hypocretin-1 in the wake-consolidated squirrel monkey. Am J Physiol Regul Integr Comp Physiol. 2007 Oct;293(4):R1736-42. doi: 10.1152/ajpregu.00460.2007. Epub 2007 Aug 8. PMID 17686881
- [Background] Zhang S, Zeitzer JM, Yoshida Y, Wisor JP, Nishino S, Edgar DM, Mignot E. Lesions of the suprachiasmatic nucleus eliminate the daily rhythm of hypocretin-1 release. Sleep. 2004 Jun 15;27(4):619-27. doi: 10.1093/sleep/27.4.619. PMID 15282996